CLINICAL TRIAL: NCT02341807
Title: A Phase 1/2 Safety Study in Subjects With CHM (Choroideremia) Gene Mutations Using an Adeno-Associated Virus Serotype 2 Vector to Deliver the Normal Human CHM Gene [AAV2-hCHM] to the Retina
Brief Title: Safety and Dose-escalation Study of AAV2-hCHM in Participants With CHM (Choroideremia) Gene Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAV2-hCHM-101
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Results first posted 2023-11-02 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Choroideremia; CHM (Choroideremia) Gene Mutations
Keywords: Choroideremia; AAV; Gene therapy; CHM; Adeno-associated virus; Adeno-associated viral vector
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: AAV2-hCHM Dose 1 (Experimental): Single, unilateral subretinal administration of a single low dose range of AAV2-hCHM.
  Interventions: Biological: AAV2-hCHM
- Cohort 2: AAV2-hCHM Dose 2 (Experimental): Single, unilateral subretinal administration of a single high dose range of AAV2-hCHM.
  Interventions: Biological: AAV2-hCHM
- Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2 (Experimental): Single, unilateral subretinal administration of a single high dose range of AAV2-hCHM.
  Interventions: Biological: AAV2-hCHM

INTERVENTIONS:
Biological: AAV2-hCHM — Comparison of different dosages of AAV2-hCHM

SUMMARY:
This clinical study evaluates the safety and tolerability of AAV2-hCHM in participants with Choroideremia gene mutations.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and tolerability of subretinal administration of AAV2-hCHM, in an inter-subject group dose escalation in individuals with choroideremia, based on a comprehensive clinical monitoring plan. The secondary objectives are to define the dose of AAV2-hCHM required to achieve stable, or improved, visual function/functional vision and to assess development of immune responses to adeno-associated virus vector, serotype 2 (AAV2) and Rab escort protein 1 (REP-1).

ELIGIBILITY:
Inclusion Criteria:

* Male at least 18 years of age diagnosed with CHM gene mutation
* Central visual field (VF) <30° in any of the 24 meridians (using Goldmann perimetry III4e isopter) in the eye to be injected
* Any evidence of functioning outer retinal cells within the central 10°

Exclusion Criteria:

* Previous history of ocular inflammatory disease (uveitis)
* Prior intraocular surgery within six months
* Participation in a previous gene therapy research trial within one year of enrollment or participation in any other ocular gene therapy trial
* Participation in a clinical study with an investigational drug in the past six months
* Grossly asymmetrical disease, or other eye morbidity, which may render the contralateral eye ineffective as a control
* Visual acuity <20/200 on standard Early Treatment of Diabetic Retinopathy Study (ETDRS) testing in the eye to be injected
* Presence of disease which may preclude the participant from participation in this trial
* Use of medications known to be neuroprotective or retino-toxic that could potentially interfere with the disease process and/or cause ocular adverse events; individuals who discontinue use of these compounds for 6 months may become eligible
* Identification by the investigator as being unable or unwilling to perform/be compliant with study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Aleman TS, Huckfeldt RM, Serrano LW, Pearson DJ, Vergilio GK, McCague S, Marshall KA, Ashtari M, Doan TM, Weigel-DiFranco CA, Biron BS, Wen XH, Chung DC, Liu E, Ferenchak K, Morgan JIW, Pierce EA, Eliott D, Bennett J, Comander J, Maguire AM. Adeno-Associated Virus Serotype 2-hCHM Subretinal Delivery to the Macula in Choroideremia: Two-Year Interim Results of an Ongoing Phase I/II Gene Therapy Trial. Ophthalmology. 2022 Oct;129(10):1177-1191. doi: 10.1016/j.ophtha.2022.06.006. Epub 2022 Jun 15. PMID 35714735

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: AAV2-hCHM Dose 1: Single, unilateral subretinal administration of a single low dose range (up to 5x10^10 vg/eye) of AAV2-hCHM (adeno-associated virus vector, serotype 2, containing the normal human choroideremia gene [CHM]).
- Cohort 2: AAV2-hCHM Dose 2; Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2: Single, unilateral subretinal administration of a single high dose range (up to 1x10^11 vg/eye) of AAV2-hCHM.
Period: Overall Study
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
Started | 5 | 5 | 5
Received at Least 1 Dose of Study Drug | 5 | 5 | 5
Completed | 5 | 4 | 5
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (7.52) | 39.6 (11.65) | 27.0 (5.00) | 34.5 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were AEs that occurred on or after the day of study drug administration. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Up to 5 years
Population: FAS included all participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
Number analyzed (Participants) | 5 | 5 | 5
Participants | 5 | 5 | 5

2. Secondary Outcome: Number of Participants With Anti-AAV2 Viral Capsid Antibody Titers That Rose Above Baseline At Least Once After Dosing
Description: Number of participants who were found to have quantifiable levels (above 1.55 micrograms [μg]/milliliter [mL]) of Anti-AAV2 viral capsid antibodies titer in the blood at least 1 study visit up to 2 years were reported.
Time Frame: Up to 2 years
Population: FAS included all participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
Number analyzed (Participants) | 5 | 5 | 5
Participants | 0 | 1 | 3

3. Secondary Outcome: Number of Participants With Cellular Immune Response to AAV2 Through Interferon Gamma Enzyme-linked Immunosorbent Spot (ELISpot) Assay
Description: Interferon gamma ELISpot assays were used to evaluate the cellular immune response to AAV2 antigen in collected peripheral blood mononuclear cell (PBMC) samples. Number of participants who demonstrated immune response to the AAV2 antigen were reported.
Time Frame: Up to 2 years
Population: FAS included all participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
Number analyzed (Participants) | 5 | 5 | 5
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Cellular Immune Response to Rab Escore Protein-1 (REP-1) Through Interferon Gamma ELISPOT Assay
Description: Interferon gamma ELISpot assays were used to evaluate the cellular immune response to REP-1 antigen in collected PBMC samples. Number of participants who demonstrated immune response to the REP-1 antigen were reported.
Time Frame: Up to 2 years
Population: FAS included all participants who received the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
Number analyzed (Participants) | 5 | 5 | 5
Participants | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: FAS included all participants who received the investigational product.
Arm/Group | Cohort 1: AAV2-hCHM Dose 1 | Cohort 2: AAV2-hCHM Dose 2 | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/5 | 2/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AAV2-hCHM Dose 1 (N=5) | Cohort 2: AAV2-hCHM Dose 2 (N=5) | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2 (N=5)
Macular hole (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extragonadal primary seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AAV2-hCHM Dose 1 (N=5) | Cohort 2: AAV2-hCHM Dose 2 (N=5) | Cohort 3 (Expansion Cohort): AAV2-hCHM Dose 2 (N=5)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 2 | 1
Cataract nuclear (Eye disorders) | 0 | 1 | 0
Cataract subcapsular (Eye disorders) | 0 | 1 | 1
Chalazion (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 4
Corneal disorder (Eye disorders) | 0 | 0 | 1
Corneal epithelium defect (Eye disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 3 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 1
Macular cyst (Eye disorders) | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Optic nerve sheath haemorrhage (Eye disorders) | 0 | 1 | 0
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1
Retinoschisis (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Visual field defect (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increase (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 1 | 0
Lymphocyte percentage abnormal (Investigations) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dellen (Eye disorders) | 1 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02341807/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02341807/SAP_001.pdf